CLINICAL TRIAL: NCT02436655
Title: Aortic Valve Replacement Versus Conservative Treatment in Asymptomatic Severe Aortic Stenosis: (AVATAR Trial): A Multicentre Randomized Controlled Trial
Brief Title: Aortic Valve Replacement Versus Conservative Treatment in Asymptomatic Severe Aortic Stenosis
Acronym: AVATAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Marko Banovic, MD PhD, FESC, FACC, Assistant Professor, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA00011929
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; normal ejection fraction; asymptomatic
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional drug treatment (No Intervention): conservative treatment and watchful waiting till symptom onset (then aortic valve replacement). Other indications for aortic valve replacement include reduced left ventricular systolic function
- elective aortic valve replacement (Active Comparator): elective aortic valve surgery (replacement) within 4 weeks after randomization
  Interventions: Procedure: surgical aortic valve replacement

INTERVENTIONS:
Procedure: surgical aortic valve replacement — open heart aortic valve replacement
  Arms: elective aortic valve replacement

SUMMARY:
Whether to intervene in asymptomatic patients with severe aortic stenosis and normal left ventricular ejection fraction remains controversial. The investigators therefore try to compare clinical outcomes of elective aortic valve replacement to conventional treatment and watchful waiting strategy in a prospective randomized trial.

DETAILED DESCRIPTION:
Aortic valve replacement (AVR) therapy is obvious choice in symptomatic severe aortic stenosis (AS) patients, because it improves symptoms, LV function and survival. Therefore, the accurate diagnosis of the disease, determination of its severity and precise evaluation of patients' clinical status is essential. However, the treatment decisions and indication for AVR in asymptomatic patients with severe AS and normal left ventricular ejection fraction (LV EF) are vague and the subject of ongoing debate. The most recent European and American guidelines have class I indication for AVR in asymptomatic severe AS patients with normal LV EF only in patients already scheduled for other cardiac surgery (for example by-pass surgery). In the case of symptom positive stress test American and European guideline differs, with European guidelines having class I indication and American guidelines only IIb indication. In all those cases of asymptomatic severe AS patients with normal LV EF the level of evidence is C, in other words there are no randomized trials. The consequence is that the decisions are made individually, patient by patient, and for this reason a patient with identical echocardiographic/clinical characteristics might be operated in USA but not in Europe (or any other part in the world), and vice-versa.

With the experience that has accumulated so far, there are retrospective and observational data that elective AVR might lead to favorable outcome compared to late (after symptom onset) surgery. This may especially come to attention with the understanding that annual risk of sudden cardiac death in asymptomatic severe AS patients with normal LV EF might be very similar or even a bit higher than operative mortality in experienced cardiac surgery centers.

Nevertheless, the majority of cardiologist worldwide are reluctant to send their asymptomatic patient with isolated severe AS and normal LV EF to AVR, and it will probably stay like that till randomized trials give us an answer whether elective AVR is beneficial.

ELIGIBILITY:
Inclusion Criteria:

* men and women of any ethnic origin aged ≥18 years
* Written informed consent
* V max across the aortic valve > 4m/s or Pmean ≥ 40mmHg and AVA ≤ 1cm2 or AVAi ≤ 0.6cm2/m2 at rest
* Without reported symptoms
* Society of Thoracic Surgeons (STS) score < 8%

Exclusion Criteria:

* Participation in another clinical trial within 30 days prior randomization
* Pregnant or nursing women
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
* Positive stress-test defined as:

  1. Anginal chest pain during testing
  2. Syncope, dizziness during testing
  3. Decrease in systolic blood pressure during exercise ≥ 20mmHg
  4. Malignant arrhythmia during exercise testing (VT or VF)
* Left ventricular ejection fraction < 50% at rest
* Very severe AS (defined as Vmax > 5.5 m/s at rest)
* Significant disease of other valves (Mitral stenosis with Pmean > 5mg, or any significant regurgitation ≥ 3+
* Recent AMI (< 1 year)
* Need for additional by-pass surgery or for aortic root replacement (i.e Bentall) or ascending aorta in asymptomatic patients undergoing AVR
* Previous by-pass surgery
* Previous any heart valve surgery
* Impaired renal function, i.e. creatinine >200 µmol/L or glomerular filtration rate < 30 mL/min/1.73 m2
* Significant pulmonary hypertension at rest (PASP > 50mmHg)
* Uncontrolled hypertension at rest (systolic >180 mmHg and diastolic >100 mmHg)
* Significant co-morbidity with reduced life expectance (< 3 years)
* Uncontrolled Diabetes Mellitus (HbA1C > 9 %)
* Significant COPD (FEV1 < 70% of predicted value)
* Permanent or paroxysmal atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
all cause death, Major Adverse Cardiac Event (MACE) including: ( Acute Myocardial Infarction - AMI, Stroke - CVI, unplanned hospitalization for Heart failure (HF) needing intravenous treatment | 36 months
all cause death, Major Adverse Cardiac Event (MACE) including: ( Acute Myocardial Infarction - AMI, Stroke - CVI, unplanned hospitalization for Heart failure (HF) needing intravenous treatment | 5 years

SECONDARY OUTCOMES:
in-hospital and 30 days operative mortality in operated patients in both groups | 30 days
repeat aortic valve surgery in operated patients in both groups | 5 years
major bleeding according to consensus report from the Bleeding Academic Research Consortium | 5 years
thromboembolic complications based on clinical symptoms, signs and imaging studies | 5 years
repeated major adverse cardiovascular events | 5 years
all-cause death + heart failure hospitalization | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marko Banovic, MD, PhD, FESC, FACC, Principal Investigator — Cardiology Department, University Clinical Centre of Serbia; Svetozar Putnik, MD, PhD, Principal Investigator — Cardiac Surgery Department, University Clinical Centre of Serbia
Locations (14):
- Cardiovascular Center Aalst, Aalst, Belgium
- Croatia (2):
  - University Clinical Center "Rebro", Zagreb
  - University Clinical Center ''Sestre milosrdnice'', Zagreb
- Czechia (2):
  - University Hospital Brno, Brno
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
- Hôpital Cardiologique de Haut Lévèque, Pessac, France
- University Hospital Galway, Galway, Ireland
- Città della Salute e della Scienza di Torino, Turin, Piedmont, Italy
- Vilnius University Hospital Santariskiu klinikos, Vilnius, Lithuania
- Medical University of Silesia, Katowice, Poland
- Serbia (4):
  - Cardiovascular Center 'Dedinje", Belgrade
  - CCSerbia, Belgrade
  - University Clinical Centre Zvezdara, Belgrade
  - Insitute for Cardiovascular Diseases "Sremska Kamenica", Novi Sad

REFERENCES:
- [Background] Banovic M, Iung B, Bartunek J, Asanin M, Beleslin B, Biocina B, Casselman F, da Costa M, Deja M, Gasparovic H, Kala P, Labrousse L, Loncar Z, Marinkovic J, Nedeljkovic I, Nedeljkovic M, Nemec P, Nikolic SD, Pencina M, Penicka M, Ristic A, Sharif F, Van Camp G, Vanderheyden M, Wojakowski W, Putnik S. Rationale and design of the Aortic Valve replAcemenT versus conservative treatment in Asymptomatic seveRe aortic stenosis (AVATAR trial): A randomized multicenter controlled event-driven trial. Am Heart J. 2016 Apr;174:147-53. doi: 10.1016/j.ahj.2016.02.001. Epub 2016 Feb 9. PMID 26995381
- [Background] Banovic M, Iung B, Bartunek J, Penicka M, Vanderheyden M, Casselman F, van Camp G, Nikolic S, Putnik S. The Aortic Valve replAcemenT versus conservative treatment in Asymptomatic seveRe aortic stenosis (AVATAR trial): A protocol update. Am Heart J. 2018 Jan;195:153-154. doi: 10.1016/j.ahj.2017.10.005. Epub 2017 Oct 14. No abstract available. PMID 29224644
- [Result] Banovic M, Putnik S, Penicka M, Doros G, Deja MA, Kockova R, Kotrc M, Glaveckaite S, Gasparovic H, Pavlovic N, Velicki L, Salizzoni S, Wojakowski W, Van Camp G, Nikolic SD, Iung B, Bartunek J; AVATAR Trial Investigators*. Aortic Valve Replacement Versus Conservative Treatment in Asymptomatic Severe Aortic Stenosis: The AVATAR Trial. Circulation. 2022 Mar;145(9):648-658. doi: 10.1161/CIRCULATIONAHA.121.057639. Epub 2021 Nov 13. PMID 34779220
- [Derived] Banovic M, Putnik S, Da Costa BR, Penicka M, Deja MA, Kotrc M, Kockova R, Glaveckaite S, Gasparovic H, Pavlovic N, Velicki L, Salizzoni S, Wojakowski W, Van Camp G, Gradinac S, Laufer M, Tomovic S, Busic I, Bojanic M, Ristic A, Klasnja A, Matkovic M, Boskovic N, Zivic K, Jovanovic M, Nikolic SD, Iung B, Bartunek J. Aortic valve replacement vs. conservative treatment in asymptomatic severe aortic stenosis: long-term follow-up of the AVATAR trial. Eur Heart J. 2024 Nov 8;45(42):4526-4535. doi: 10.1093/eurheartj/ehae585. PMID 39217448
- [Derived] Zelis JM, Tonino PAL, Pijls NHJ, De Bruyne B, Kirkeeide RL, Gould KL, Johnson NP. Coronary Microcirculation in Aortic Stenosis: Pathophysiology, Invasive Assessment, and Future Directions. J Interv Cardiol. 2020 Jul 22;2020:4603169. doi: 10.1155/2020/4603169. eCollection 2020. PMID 32774184

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02436655/SAP_000.pdf